CLINICAL TRIAL: NCT00859261
Title: 2D Silicon Transducer-Compression Plates for Breast Ultrasound
Brief Title: Two Dimensional (2D) Silicon Transducer-Compression Plates for Breast Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul L. Carson Ph.D, Principal Investigator ( Ph.D ), University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HUM 15464; 2R01CA091713 (NIH); R01CA115267 (NIH)
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Breast Tumor; Breast Cysts
MeSH Terms: conditions — Breast Neoplasms; Breast Cyst

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Breast imaging using Ultrasound and Photoacoustic (Experimental): Evaluating 3D ultrasound for breast abnormalities/masses/cysts. This includes ultrasound imaging and possibly photoacoustic imaging.
  Interventions: Procedure: Experimental 3D Breast Ultrasound imaging; Procedure: Experimental Photoacoustic Imaging

INTERVENTIONS:
Procedure: Experimental 3D Breast Ultrasound imaging — Subjects will be seated and have the indicated breast positioned in the 3D breast ultrasound imaging device. An ultrasound gel will be applied to the breast by the technician. The breast will be gently compressed between the ultrasound plates to facilitate the 3D (dimensional)breast imaging. This imaging session will take approximately 30 minutes to complete.
Procedure: Experimental Photoacoustic Imaging — Subjects will be placed in a seated position for the photoacoustic tomography(PAT) imaging. The subjects will be given a laser protective mask to wear. Each subject will be instructed how to wear this mask(goggles) to protect their eyes during the imaging session. Pulse monitor leads may be placed on their chest to allow the computer to record the images of blood flow in the breast. The breast will be placed on the laser device platform and positioned so that the laser beam is appropriately directed to the targeted area of the breast. During the imaging the temperature of the skin under laser light, will be checked often with a thermometer to make sure that the skin is not getting too hot. This laser based imaging scan will take approximately 10 minutes to complete.
  Other Names: Photoacoustic Tomography (PAT)

SUMMARY:
The study purpose is to help in the developement of 3 dimensional breast ultrasound imaging.

DETAILED DESCRIPTION:
To assist in the developement of 3 dimensional breast ultrasound imaging and when possible compare the ultrasound results with 3D mammography (digital tomosynthesis mammography)or clinical mammography and ultrasound. Hopefully that this new, 3D ultrasound imaging can provide important information not found on mammograms or routine breast ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women OR
* Women with suspected benign masses who may/or may not be going to biopsy
* Women with cysts where no biopsy is recommended

Exclusion Criteria:

* Women who are pregnant
* Women with breast implants
* Prisoners

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To prove the significance/capability of 3D Ultrasound imaging in comparison to current mammographic imaging. | 1 year
  Assess the quality of 3 D ultrasound in comparison to conventional mammography

CONTACTS AND LOCATIONS:
Overall Officials: Paul Carson, Ph.D., Principal Investigator — University of Michigan Basic Science Division
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No